CLINICAL TRIAL: NCT03003897
Title: Effects of Soluble Fiber Consumption on Body Weight, Glycemia, and Insulinemia in Adults With Overweight and Obesity: a Systematic Review and Meta-analysis of Randomized Controlled Trials.
Brief Title: Meta-analysis of Soluble Fiber Consumption on Body Weight, Glycemia, and Insulinemia in Overweight and Obese Adults.
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Other Study IDs: Soluble Fiber Review
Record Dates: First submitted 2016-10-28; First posted 2016-12-28 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: Dietary Fiber; Soluble Fiber; Body Mass Index; Body Weight; Blood Glucose; Insulin
MeSH Terms: conditions — Obesity; Body Weight; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Soluble Fiber Treatment: Participants receiving soluble fiber.
  Interventions: Other: Soluble Fiber
- Placebo Treatment: Participants receiving placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Soluble Fiber — Participants receiving soluble fiber.
  Groups: Soluble Fiber Treatment
Other: Placebo — Participants receiving placebo.
  Groups: Placebo Treatment

SUMMARY:
Dietary fiber intake is protective against overweight and obesity; however, a significant fiber gap exists between consumption and recommended intake values. Soluble fiber beneficially impacts metabolism, and supplementation may be a feasible approach to improve body composition and glycemia in overweight and obese individuals. The investigators will evaluate results of randomized controlled trials (RCTs) of soluble fiber supplementation among overweight and obese adults for outcomes related to weight management (e.g. body mass index [BMI], body weight, body fat percentage, waist circumference) and glucose and insulin homeostasis (e.g. fasting glucose, homeostasis model assessment of insulin resistance [HOMA-IR], fasting insulin) through systematic review and meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

Peer-reviewed randomized controlled trials (RCTs) will be included in the systematic review and meta-analysis if they involve participants who are:

1. Overweight or obese (BMI ≥ 25.0 kg/m2 for U.S. populations and ≥ 23.0 kg/m2 for Asian populations and/or waist circumference ≥ 40 inches (94 cm) in men or ≥ 35 inches (80 cm) in women and/or waist-to-hip ratio ≥ 0.90 in men or ≥ 0.85 in women).
2. Weight stable and not actively trying to lose weight at screening.
3. Without physician-diagnosed chronic conditions at screening (e.g., dyslipidemia, hypertension, type 2 diabetes, and cardiovascular disease).
4. Included studies will be soluble fiber supplementation interventions that are controlled feeding studies or conducted among free-living subjects that provide data for outcomes of interest.

Exclusion Criteria:

Studies will be excluded from the systematic review and meta-analysis if they meet any of the following criteria:

1. Studies conducted in animals.
2. Mechanistic research.
3. Human trials involving pregnant women, breastfeeding women, or children.
4. Conference proceedings.
5. Articles not published in English.
6. Studies less than 1 week in duration.
7. Studies that pool outcome measure data for healthy weight and overweight and obese individuals.
8. Studies involving whole food treatments or high fiber profile diets.
9. Weight loss interventions involving other tactics, such as counseling or energy restriction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥ 18 years of age with overweight and obesity but without physician diagnosed chronic disease at screening.
Sampling Method: Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Body mass index (kg/m2) | ≥ 1 week
Body weight (kg) | ≥ 1 week
Body fat (% fat mass) | ≥ 1 week
Waist circumference (cm) | ≥ 1 week
Fasting glucose (mmol/l) | ≥ 1 week
Fasting insulin (pmol/l) | ≥ 1 week
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | ≥ 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data has been previously published in the randomized controlled trials we intend to analyze.

REFERENCES:
- [Result] Thompson SV, Hannon BA, An R, Holscher HD. Effects of isolated soluble fiber supplementation on body weight, glycemia, and insulinemia in adults with overweight and obesity: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2017 Dec;106(6):1514-1528. doi: 10.3945/ajcn.117.163246. Epub 2017 Nov 1. PMID 29092878